CLINICAL TRIAL: NCT05767372
Title: Effect of Coherent Breathing on Different Outcome Measures in Elderly
Brief Title: Effect of Coherent Breathing on Elderly Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Elbanna, lecturer at faculty of physical therapy at Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dr Sherif Elabd
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Stable Diabetes Mellitus; Geriatrics; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coherent breathing group (Experimental): The participants will receive Inspiratory muscle trainer and Coherent breathing exercise three times per week for 12 weeks.
  Interventions: Other: Coherent Breathing Exercise
- Inspiratory muscle training group (Experimental): The participants will receive Inspiratory muscle training three times per week for 12 weeks.
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Other: Coherent Breathing Exercise — Step 1: Focus on your natural breathing and count the time of your inhale and exhale.
  Step 2: Sit in a comfortable position to practice the coherent breathing technique. Gently place one hand on your stomach.
  Step 3: Inhale for four seconds and then exhale for four seconds. Repeat this for one minute.
  Step 4: Repeat the above step but lengthen your inhales and exhale for five seconds.
  Step 5: Repeat the above step but extend the breaths to six seconds. Once you're able to do this for five minutes, gradually work your way up to 20 minutes.
  During this breathing exercise, keep your hand on your stomach. Using diaphragmatic breathing can help you feel your breaths.
  Arms: Coherent breathing group
Device: Inspiratory muscle training — The patient was in the comfortable sitting position and then put the nose clip on the patient's nose
  1. After setting the maximum training; the user recognized the load at which they could effectively execute ten breaths at greatest resistance relying upon the patient's pace of apparent effort.
  2. Training was begun with a load at low intensity 20-30% of the patient maximum 10 repetition method using inspiratory muscle training (IMT) device.
  3. Progress slowly and monitor carefully.
  4. As the inspiratory muscle became stronger the inspiratory load was progressed to 50% of maximum effort over 3 weeks as tolerated.
  5. Patient took full breath in (maximal and deep inspiration) then longer and slow expiration. Continue this breathing pattern for 10-20 breath.
  6. Repeated step (5), 4-6 times or about 10-15minutes with rest in between 30 seconds.
  7. The session was repeated three times per week for 12 weeks.
  Arms: Inspiratory muscle training group

SUMMARY:
This study will be carried out on sixty elderlies of both gender with ages ranges from 60 to 70 years old. The participants will receive Inspiratory muscle trainer and/or Coherent breathing exercise three times per week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly subject of both gender with age ranged from 60 to 70 years old.
2. BMI will be ranged from 25 to 29.9.
3. Clinically and medically stable.
4. Able to understand the requirements of the study.
5. Conscious patient and respond to verbal command.

Exclusion Criteria:

1. Neurological conditions (e.g., stroke history, Parkinson's disease).
2. Presence of an acute illness.
3. Metabolically unstable chronic illness.
4. Pre-existent untreated metabolic or renal disease.
5. Patient undergoes chemotherapy.
6. Recent surgery.
7. Uncontrolled diabetes or hypertension.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Tinetti Performance Oriented Mobility Assessment (POMA) | 12 weeks
  Evaluating tests of balance and gait
  Description:
  The Tinetti assessment tool is an easily administered task-oriented test that measures an older adult's Scoring: A three-point ordinal scale, ranging from 0-2. "0" indicates the highest level of impairment and "2" the individuals independence. Total Balance Score = 16 Total Gait Score = 12 Total Test Score = 28 Interpretation: 25-28 = low fall risk 19-24 = medium fall risk < 19 = high fall risk
The five Times Sit to Stand Test | 12 weeks
  Evaluating fall risk
The muscle quality index (MQI) | 12 weeks
  Evaluating age-related alterations in muscle function
The Geriatric Depression Scale (GDS) | 12 weeks
  Evaluating psychological aspect Of the 15 items, 10 indicated the presence of depression when answered positively, while the rest (question numbers 1, 5, 7, 11, 13) indicated depression when answered negatively. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
The 6 minutes' walk test (6MWT) | 12 weeks
  Evaluating aerobic fitness
Short form Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) | 12 weeks
  Evaluating cognitive decline
  * Minimum score: 16
  * Maximum score: 80
  * High score means worse outcome.
Evaluation of oxygen saturation (SPO2) and heart rate (HR) | 12 weeks
  By using the pulse oximeter.

SECONDARY OUTCOMES:
Modified Borg Dyspnoea Scale | 12 weeks
  Evaluating level of exertion during exercise It starts at number 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal
Evaluation of forced expiratory volume at one second (FEV1) and maximum voluntary ventilation (MVV) | 12 weeks
  By using spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Sherif O Elabd, Master, Principal Investigator — May University
Locations (1):
- Faculty of physical therapy outpatient clinic, Cairo, Giza Governorate, Egypt